CLINICAL TRIAL: NCT05651763
Title: The Effects of Transcranial Direct Current Stimulation Associated With Pilates Based Exercise in Performance of Patients With Chronic Low Back Pain
Brief Title: Transcranial Direct Current Stimulation Associated With Pilates in Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRAG2022
Record Dates: First submitted 2022-12-06; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain; Transcranial Direct Current Stimulation
Keywords: Transcranial Direct Current Stimulation; Low back pain; Exercises; Chronic pain; Performance; Treatment
MeSH Terms: conditions — Low Back Pain; Motor Activity; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation and exercise group (Experimental): 30-minute exercise program (based on Pilates method) associated with active transcranial direct current stimulation.
  Interventions: Other: Stimulation and exercise group
- Exercise and sham stimulation group (Sham Comparator): 30-minute exercise program (based on Pilates method) associated with sham transcranial direct current stimulation.
  Interventions: Other: Exercise and sham stimulation group

INTERVENTIONS:
Other: Stimulation and exercise group — Exercise protocol + application of active direct current stimulation for 30 minutes.
  Arms: Stimulation and exercise group
Other: Exercise and sham stimulation group — Sham Transcranial direct current stimulation Exercise protocol + application of simulation of direct current stimulation for 30 minutes. The stimulator will be turned off after 30 seconds and the volunteers will not receive current for the rest of the session.
  Arms: Exercise and sham stimulation group

SUMMARY:
This is a randomized and blind clinical trial, whose objective is to evaluate the effects of transcranial stimulation by direct current associated with exercises based on the pilates method on the performance of patients with chronic low back pain.

DETAILED DESCRIPTION:
Considered a public health problem, low back pain is globally presented as a symptomatology of high prevalence, incidence and recurrence. In addition, it is responsible for a large part of disabilities, reduced functional performance, absences from work and impaired quality of life, which brings biopsychosocial impacts to the affected subjects. Treatments that relieve the symptoms of these patients are of great importance to improve the quality of life of these individuals. Thus, this study aims to evaluate the effects of transcranial direct current stimulation associated with Pilates based exercise on chronic low back pain. This is a randomized clinical trial that will be composed of women between 18 and 65 years of age, with a history of low back pain for more than 12 weeks and a minimum pain intensity equal to 3 cm on the numerical pain scale. The volunteers will be randomized into two distinct groups: stimulation + exercise group (EG - will perform a Pilates based exercise protocol combined with transcranial direct current stimulation) and sham stimulation + exercise group (SG - will perform the same exercise program combined with sham stimulation). The interventions, regardless of the group, will be carried out three times a week for four weeks. Participants will be submitted to three assessments: the first (T0) will be performed before the treatment protocols; the second (T1) will be performed after the four weeks of intervention; and the third (T2) will be a follow-up one month after the end of the treatment protocol. Pain sensation, performance, pressure pain threshold, use will be evaluated. For the statistical analysis, a mixed model ANOVA will be performed for the inter and intragroup comparison, with Tukey's post hoc, considering a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

Women with chronic nonspecific low back pain (for more than 12 weeks) and minimum pain intensity of 3 on numerical pain rating scale

Exclusion Criteria:

* diagnosis of fracture and spine pathologies, fibromyalgia, spine surgery in the last year;
* low cognitive level assessed by the Mini Mental State Examination;
* presence of central neurological diseases (such as Parkinson's and stroke) or psychiatric (such as depression or schizophrenia);
* history of epileptic illness;
* seizure history;
* brain implants;
* pacemaker;
* pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (numerical pain rating scale) | up to 1 month of follow-up
  Pain intensity measured by numerical pain rating scale, measured on an 11-point where 0=no pain and 10=worst possible pain.

SECONDARY OUTCOMES:
Pressure pain threshold | A pressure pain four weeks after intervention and 1 month of follow-up
  Pressure pain threshold measured by pressure algometer.
Root Mean Square (RMS) | Evaluation of RMS four weeks after intervention and 1 month of follow-up
  Analyze of the electromyographic activity of the back muscles
Peak of muscular torque | Evaluation of Peak of muscular torque four weeks after intervention and 1 month of follow-up
  Evaluate the peak of muscular torque using the hand-held dynamometer.
Back muscle fatigue | Evaluation of Back muscle fatigue four weeks after intervention and 1 month of follow-up
  Measure the back muscular resistance to fatigue using the Ito test

IPD SHARING:
Plan to Share IPD: No